CLINICAL TRIAL: NCT03435120
Title: Quality of Life Study in Patients With Breakthrough Cancer Pain Treated in Medical Oncology Services
Brief Title: Quality of Life Study Breakthrough Cancer Pain Treated in Medical Oncology Services (CAVIDIOM)
Acronym: CAVIDIOM
Status: Completed | Type: Observational
Sponsor: Angelini Farmacéutica (Industry)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: ANG-ANA-2017-01 (CAVIDIOM)
Record Dates: First submitted 2018-01-29; First posted 2018-02-15 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Breakthrough Pain
Keywords: Breakthrough Cancer Pain; Quality of life; Medical Oncology
MeSH Terms: conditions — Breakthrough Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breakthrough Cancer Pain: No intervention (Non Interventional Study)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In cancer patients, pain is one of the most common symptoms. The range of reported prevalence of pain varies from 33% to 64% including different stages of cancer, during or after anticancer treatment. Moreover, despite the optimal management of basal chronic pain, 66% of these patients have reported breakthrough pain which has a severe impact on quality of life. There is insufficient clinical information on the quality of life of cancer patients with breakthrough pain treated in medical oncology services according to routine clinical practice. For this reason we consider it is appropriate to prospectively evaluate the quality of life of cancer patients with cancer breakthrough pain in medical oncology services as well as other factors that can affect quality of life. This post-authorization observational study will assess the quality of life of cancer patients with breakthrough cancer pain treated in medical oncology services in Spanish hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Patients with histologically confirmed neoplasia
* Patients attended in medical oncology consultations
* Life expectancy > 3 months
* Patients with baseline controlled cancer pain with opioids who are diagnosed of breakthrough cancer pain by Davies algorithm
* Written informed consent

Exclusion Criteria:

* Untreated patients with opioids for baseline pain
* Patients who are not opioid tolerant
* Serious psychiatric disorder or any disease or condition that prevents the collection of data
* Patients with evidence of opioid addiction or history of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breakthrough cancer pain treated in Medical Oncology services
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Changes in quality of life of the patients | Up to 4 weeks
  Changes according to EQ-5D-5L questionnaire

SECONDARY OUTCOMES:
Characteristics of patients | At baseline
  Kind of tumor.
Characteristics of patients | At baseline
  Demographic data
Characteristics of patients | At baseline
  ECOG
Management of cancer breakthrough pain. | Up to 4 weeks
  Cancer breakthrough pain characteristics (time until maximum intensity)
Management of cancer breakthrough pain. | Up to 4 weeks
  Cancer breakthrough pain evolution (duration and management)
Anxiety and depression status and the possible relationship between these factors and quality of life. | Up to 4 weeks
  Goldberg Anxiety and Depression Scale.
Sleep quality and the possible relationship between this factor and quality of life. | Up to 4 weeks
  MOS sleep questionnaire
Evaluate caregivers effort | Up to 4 weeks
  Results according to caregivers effort Index
Perceived assistance quality by patients | Up to 4 weeks
  Results according to Sociofamily evaluation scale of "Gijon"
Improvement impression perceived by patients | Up to 4 weeks
  Results according to assessment of perceived quality (questionnaire of the Ministry of Health and Consumer Affairs)
Improvement impression perceived by patients | Up to 4 weeks
  Results according to Satisfaction questionnaire PGI-I
Improvement impression perceived by patients | Up to 4 weeks
  Results according to Satisfaction questionnaire CGI-I

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Camps Herrero, Principal Investigator — Hospital General Universitario de Valencia
Locations (14):
- Spain (14):
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca, Palma
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitari de San Joan de Reus, Reus, Tarragona
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Universitario La Paz, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Alvaro Cunqueiro, Vigo
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No